CLINICAL TRIAL: NCT06627738
Title: Locally Advanced NSCLC Treated With Radiochemotherapy: Phase 2 Study on the Value of a Stereotactic Boost
Acronym: Cybertaxcis II
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022/17; 2024-A01394-43 (Other: ANSM)
Record Dates: First submitted 2024-10-03; First posted 2024-10-04 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arms (Experimental): After their radiochemotherpy (Taxcis protocol), the eligible patients will be included in the study and will have a Cyberknife boost (5 sessions of 8 Gray, over 2 weeks maximum). They will have follow-up visits for 2 years post-treatment. Then, their disease and survival status will be recorded until 5 years post-treatment.
  Interventions: Radiation: Cyberknife irradiation

INTERVENTIONS:
Radiation: Cyberknife irradiation — Additional Cyberknife irradiation after a doublet of Platinum Salts-based chemotherapy and concomitant radiotherapy in inoperable patients with locally advanced non-small cell lung carcinoma

SUMMARY:
This is a monocentric, non-randomized, open-label, superiority phase II clinical investigation evaluating the efficacy of additional Cyberknife irradiation after a doublet of Platinum Salts-based chemotherapy and concomitant radiotherapy in patients with locally advanced non-small cell lung carcinoma (NSCLC), with an interim analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years old or more
2. ECOG 0 to 2
3. Histologically proven non-small cell lung cancer
4. Stage III non-metastatic tumor, not allowing for immediate surgery
5. Volume(s) on the evaluation chest CT scan done at the end of conventional radiotherapy (between 34 & 46 Gy) meeting the following criteria:

   * 1 to 3 target volumes of less than 5 cm in greatest diameter
   * And allowing for the delivery of a CyberKnife boost to be carried out in compliance with the manufacturer requirements and with the doses delivered to the organs at risk (OAR/fractions) defined in appendix 2
6. Patients who have received a " Taxcis " treatment consisting in 2 cycles of induction chemotherapy (platinium-based doublet) and then at least 40 Gy of irradiation in combination with at least 2 cycles of concomitant chemotherapy (platinium-based doublet)
7. No contraindication to implantable venous devices (IVDs)
8. Patient who has read the patient information note and signed the consent form
9. If applicable, negative pregnancy test*
10. Eligible for National Health Insurance in France
11. Chest CT scan performed prior to Taxcis

Exclusion Criteria:

1. Positive EGFR mutation
2. Exercise-induced dyspnea associated with heart failure equal to or greater than stage III of the New York Heart Association (NYHA) classification, (appendix 3)
3. Coronary syndrome or heart failure in the last three months
4. Pulmonary function test contraindicating radiotherapy: PFT-FEV1 inferior to 1 L.
5. After radio-chemotherapy, presence of any toxicity contraindicating Cyberknife irradiation
6. Vulnerable populations and participants as defined in Articles 64 to 68 of Regulation (EU) 2017/745 of the European Parliament and of the Council of 5 April 2017:

   * Incapacitated participants who have not given or refused informed consent prior to the onset of their incapacity, who are not under the provisions of article 64 ;
   * Pregnant or breast-feeding women who are not covered by the provisions of article 66 ;
   * Adults under legal protection or unable to express their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2034-02 (Estimated); Study Completion 2034-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate progression-free survival at 24 months after additional Cyberknife irradiation following concomitant radio-chemotherapy in patients with locally advanced non-small cell lung carcinoma (NSCLC). | 24 months
  Progression-free survival at 24 months will be assessed by calculating the time between the date of inclusion and the date of progression (according to RECIST 1.1 criteria) or death from any cause whichever come first. Patients who have not progressed, died or been lost to follow-up at the time of analysis will be censored at the date of last news.

SECONDARY OUTCOMES:
Evaluate overall survival at 24 months and at 60 months | 60 months
  Overall survival at 24 months and at 60 months will be assessed by calculating the time between the date of inclusion and the date of death from all causes. Patients who have not died or been lost to follow-up at the time of analysis will be censored at the date of last news.
Evaluate specific survival at 24 months and at 60 months | 60 months
  Specific survival at 24 months and at 60 months will be assessed by calculating the time between the inclusion and the date of cancer-related death. Patients who have not died or been lost to follow-up at the time of analysis will be censored at the date of last news.
Evaluate the efficacy of the additional Cyberknife irradiation following concomitant radio-chemotherapy at 24 months | 24 months
  The overall response rate (complete or partial response, stabilization, progression) at 24 months will be defined by RECIST v 1.1 criteria. The objective response rate (CR or PR) will be estimated as the number of patients with a documented complete or partial response, divided by the number of analyzable patients, described for each evaluation. The median duration of response will be given with its 95% confidence interval.
Evaluate overall tolerability of the additional Cyberknife irradiation following concomitant radio-chemotherapy at 24 months | 24 months
  The overall tolerability of the additional Cyberknife irradiation following concomitant radio-chemotherapy throughout patient participation will be evaluated by clinical and biological means and rated according to the NCI CTCAE V5.0 scale.
Evaluate overall quality of life before Cyberknife, 1 month post-Cyberknife and 6 months post-Cyberknife | 6 months
  Quality of life will be assessed using the EORTC QLQ-C30 questionnaire (items 29-30)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Antoine Lacassagne, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided